CLINICAL TRIAL: NCT05112510
Title: Prognostic Prediction of Nasopharyngeal Carcinoma Based on Radiomics Features of MR Diffusion-weighted Imaging
Brief Title: Prognostic Prediction of NPC Based on MR Diffusion-weighted Imaging
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: ZDWY.HYXK.003
Record Dates: First submitted 2021-10-17; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Patients With Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- event group: The patients with nasopharyngeal carcinoma developed distant metastasis or recurrence after standard treatment.
  Interventions: Other: Observing whether developing distant metastasis or recurrence
- non-event group: The patients with nasopharyngeal carcinoma did not develop distant metastasis or recurrence after standard treatment.
  Interventions: Other: Observing whether developing distant metastasis or recurrence

INTERVENTIONS:
Other: Observing whether developing distant metastasis or recurrence — The study is a observational study and has no intervention.

SUMMARY:
The purpose of this study is to explore whether the imaging model based on RESOLVE-DWI sequence can exploiting the heterogeneity of nasopharyngeal carcinoma and indicate the prognosis, so as to provide intervention information for clinical decision-making. All patients were randomly divided into the training group and the validation group. Radiomics features extracted from T2-weighted, DWI, apparent diffusion coefficient (ADC), and contrast- enhanced T1-weighted were used to build a radiomics model. Patients'clinical variables were also obtained to build a clinical model. Model of training cohort was established using cross-validation for nasopharyngeal carcinoma prognosis by machine learning, including Logistics Regression, SVM, KNN, Decision Tree, Random Forest, XGBoost, and then, the model will be verified in the validation cohort. Area under the curve (AUC) of the Machine learning model was used as the main evaluation metric.

ELIGIBILITY:
Inclusion Criteria:

1. patients with nasopharyngeal carcinoma diagnosed by pathology;
2. complete clinical data and MR imaging data;
3. without radiotherapy, chemotherapy or operation before MR examination.

Exclusion Criteria:

1. incomplete follow-up data;
2. poor image quality and can not be used for analysis;
3. patients with other tumors in the past or at the same time.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient with nasopharyngeal carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Calculating AUC of machine learning model based on MR diffusion-weighted imaging to evaluate efficacy for prognosis | Before January 2022
  After building machine learning model based on the features extracted by MR diffusion-weighted imaging of patients with nasopharyngeal carcinoma. Some measurements will be output from machine learning model such as AUC、F1、Accuracy and so on. Area under the curve (AUC) of the Machine learning model will be used as the main evaluation metric to evaluate the efficacy of a machine learning model which is used to predict the prognosis of patients with nasopharyngeal carcinoma (NPC).

SECONDARY OUTCOMES:
Comparing AUC of machine learning model based on MR diffusion-weighted imaging and conventional MR sequences for prognosis | Before January 2022
  After separately building machine learning model based on the highly correlated features extracted by MR diffusion-weighted imaging and conventional MR sequences of patients with nasopharyngeal carcinoma. Some measurements will be output from the machine learning models such as AUC、F1、Accuracy and so on. Area under the curve (AUC) of the Machine learning model will be used as the main evaluation metric to study if the prediction efficiency of the machine learning model based on the highly correlated features extracted by MR diffusion weighted imaging imaging is better than that of conventional MR sequences.
Calculating AUC of machine learning model based on MR diffusion-weighted imaging combinated with conventional MR sequence to evaluate efficacy for prognosis | Before January 2022
  Fianlly, we build a machine learning model based on MR diffusion-weighted imaging combinated with conventional MR sequences from patients with nasopharyngeal carcinoma. Some measurements will be output from the machine learning models such as AUC、F1、Accuracy and so on. Area under the curve (AUC) of the Machine learning model will be used as the main evaluation metric to explore whether the machine learning model established by imaging features of MR diffusion-weighted imaging and conventional MR sequence has best prediction efficiency comparing with the models mentioned above.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China